CLINICAL TRIAL: NCT06820879
Title: Viscoelastic Tests (VET) Versus Conventional Coagulation Tests (CCT) for Management of Trauma-Induced Coagulopathy: Opened, Randomized, Two-Parallel, Controlled Trial.VISCOTAC
Brief Title: Viscoelastic Tests (VET) Versus Conventional Coagulation Tests (CCT) for Management of Trauma-Induced Coagulopathy
Acronym: VISCOTAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0937
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Trauma Coagulopathy
Keywords: Coagulopathy; coagulation tests; viscoelastic tests; massives transfusions; labile blood products
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional arm: conventional coagulation tests. (No Intervention): In this arm, patients will have a detection and a correction of the TIC based on conventional coagulation assays. The threshold used to initiate a correction, in case of ongoing bleeding, will be set at fibrinogen concentration ≤ 1.5 gr/L, PTratio >1.5 or platelets < 50 G.L-1 (< 100 G.L-1 in case of severe brain injury).
- Viscoelastic arm: Viscoelastic Tests (Experimental): The detection and correction of TIC will be based on viscoelastic assay using values of clotting time (CT EXTEM), clot amplitude at 5 minutes (A5 FIBTEM and A5 EXTEM) and maximum lysis (ML). The algorithm for the study has been recently published and is based on thresholds for EXTEM (CT, A5 and ML), FIBTEM (A5). The algorithmic correction by fibrinogen concentrates and FFP is initiated using different cutoffs and parameters than in control arm, but the quantity of fibrinogen concentrates and FFP transfused will be similar in both arms.
  Interventions: Device: Viscoelastic Tests (ROTEM)

INTERVENTIONS:
Device: Viscoelastic Tests (ROTEM) — Viscoelastic Tests (2-6 tests for the study over the first 24 hours)
  Arms: Viscoelastic arm: Viscoelastic Tests

SUMMARY:
Traumatic coagulopathy is a complex, multifactorial event that occurs in 20-30% of patients on admission. It increases mortality, and its treatment is one of the main priorities in the early management of severely injured patients. Diagnosis of coagulopathy has traditionally been based on conventional coagulation tests (CCTs), which provide an assessment of patients' coagulation in over 60 minutes. Over the past fifteen years, viscoelastic tests (VETs) have been proposed, providing a more rapid result (≤ 10 min) and can guide the administration of labile blood products (LBP). Various studies, mainly retrospective, have shown that the use of VETs is associated with a significant reduction in the use of LBP and the incidence of massive transfusions (MT).

For example, it has been showed that the use of VETs was accompanied by a reduction in the administration of LBP and more particularly of RBC (Red blood cell concentrate) (4.8 units vs. 1.9 units). The investigators obtained the same result on a larger number of patients, with a further reduction in the administration of other LBP and in the incidence of MT (33% vs. 8%, p<0.01).

However, the main limitation of these 2 studies is that the results may not have been due solely to the use of ROTEM, but rather to a care package combining the use of ROTEM with the administration of tranexamic acid and the implementation of Damage Control Surgery techniques.

To avoid this methodological criticism, we recently compared 2 contemporary French cohorts (2012-2019), in which patients had similar management of traumatic injuries, with the exception of the type of coagulation tests: CCT vs. VET. The use of VET s was associated with an increase in the number of patients alive at 24h without MT (76% vs. 55%, p<0.001), but also with a sharp reduction in the administration of all LBPs.

This composite criterion associating the occurrence of a MT with survival at 24 hours after hospital admission was the primary endpoint of the randomized iTACTIC study. iTACTICS was published in 2021, and aimed to compare in severely injured patients 2 strategies for the diagnosis and treatment of coagulopathies, based on CCT in one arm and VET in the other. In this work, the use of VET was not associated with an improvement in the proportion of patients alive at 24 hours without MT (64% vs. 67%, OR 1.15, CI95%: 0.8-1.7), nor with any of the other criteria studied. The main limitation of this study is that less than a third of the patients included had a coagulopathy on admission. The probability of receiving LBP was therefore low. In the subgroup of the most severe patients, an improvement in the primary endpoint was observed for patients randomized to the VET group. The small sample size and subgroup analysis, however, limited the significance of this result.

All these elements suggest that it is necessary :

* to use a composite endpoint rather than a single endpoint (mortality) for the evaluation of VET-based strategies, combining early mortality with the occurrence of a transfusion event.
* conduct a randomized trial comparing the use of VETs with that of CCTs in trauma patients with a high probability of coagulopathy on admission to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Blunt or penetrating injury
* Less than 3 hours after a trauma AND less than 1 hour after trauma room admission
* One of the following criteria:

  * Severe trauma in shock (shock index > 0.9 or SBP < 90 mmHg) or with anemia (hemoglobin < 11 g.dL-1) and at least 1 of the following criteria:

    * Positive extended-FAST (Focused Assessment with Sonography for Trauma, ultrasound) finding liquid
    * Severe bone injury :

      * Fracture of at least two long bones
      * Amputation above the knee or elbow
    * Open fracture of the pelvis and/or mechanically unstable pelvis
  * Severe trauma with a high probability of having a TIC (PTratio > 1.20) according to the TIC score (score value ≥ 6 - cf. appendix 2)
* Emergency procedure with secondary informed consent signed by the patient

Exclusion Criteria:

* Known pregnancy at admission
* Transfer from another hospital
* Cardiac arrest before randomization
* Patient with devastating injuries expected to die within the first hour post-admission
* Massive head injury with GCS 3 and bilateral mydriasis
* Pre-hospital transfusion of RBCs unit or coagulation factors concentrates
* No tranexamic acid before hospital admission
* Patient with uncontrolled major bleeding on arrival with direct admission to the operating room for rescue surgery
* Conventional or viscoelastic assay before inclusion/randomization
* Hypothermia < 33°C
* Known use of oral anticoagulants (VKA or DOACs)
* Known congenital hemostasis abnormality
* Predictable transfer to another hospital <12 hours after admission
* Patients protected by articles L1121-6 and L1121-7 of the Public Health Code, adults subject to legal protection measures
* Patient not affiliated to a social security scheme
* Patient included in other interventional study on coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The survival without massive transfusion 24 hours after admission in the VET arm as compared to the CCT arm. | 24hours after admission
  24 hours after admission in the VET arm as compared to the CCT arm. The survival 24 hours after admission will be combine with the non-occurrence of massive transfusion (i.e., at least 10 units of RBC received at 24h).
  This comparison will be first carried out in a crude manner, and then considering the stratification factor, i.e., a Glasgow Coma Scale < 9 (severe traumatic brain injury) and administration of plasma (FFP or lyophilized plasma).

SECONDARY OUTCOMES:
Number and proportion of patient receiving labile blood products, at 4, 6 and 24 hours after hospital admission. | 4, 6 and 24 hours after hospital admission
Number and proportion of patients receiving fibrinogen concentrates as well as the quantity administered (in grams), at 6 and 24 hours after hospital admission | 6 and 24 hours after hospital admission
Number and proportion of patients who received massive transfusion, time critical transfusion and Rescue therapy | 24 hours
  * A massive transfusion (MT, ≥ 10 RBC at H24)
  * A time critical transfusion (≥ 6 RBC at H6 following the admission).
  * Rescue therapy, defined as the emergency administration of blood products because the patient's clinical condition makes it impossible to wait for the results of biological tests (CCT or VTE).
Number of RBCs received from admission to ICU discharge (or at 28 days maximum after randomization (Day 28)). | At discharge or at 28 days maximum after randomization (Day 28))
Number and proportion of patients with a "Sepsis-related Organ Failure Assessment" (SOFA) score > 5, after randomization, at H24, Day 2, Day 3, Day 4. | 4 days
Ventilator-free days, vasopressor days, renal replacement therapy days | 28 days
  Ventilator-free days (Calculated by the subtracting the number of days spent on mechanical ventilation from 28), vasopressor days (calculated as the total number of days spent on inotropic drugs, for example noradrenaline), renal replacement therapy days (calculated as the total number of days spent on hemofiltration or hemodialysis).
Total volume (mL) of fluids received at 24-hours including blood products and fluid resuscitation (crystalloids and colloids). | H24
Number and proportion of patients who died at H6, H24 and Day 28 | 28 days
  * For any reason (crude mortality)
  * By ISS score value (9-15=moderate trauma, 16-24 = severe trauma, ≥ 25 = very severe trauma) and stratified on the occurrence of brain-injury (defined by head AIS > 3), according to shock define by a lactate more than 3.9 mmol.l-1
  * By attributable cause of death, including trauma brain injuries, bleeding, anoxia, sepsis, other The time median between randomization and the occurrence of death will be measured and compared between trial arms.
Length of stay in the intensive care unit up to Day 28. | 28 days
Timing and the number of hemorrhage control procedures (surgery, interventional radiology) in the first 6-hours following admission. | 6 hours
Number and proportion of patients with grade 3 and 4 adverse events related to the management strategy between randomization and Day 28 | 28 days
  * Ventilator-associated pneumonia
  * Acute Respiratory Distress Syndrome (ARDS)
  * Acute renal failure as defined by KDIGO (Kidney Disease / Improving Global Outcome 2012)
  * Septic shock defined
  * Any thromboembolic event; pulmonary embolism, deep vein thrombosis, gastrointestinal ischemia, non-traumatic limb ischemia, myocardial infarction, ischemic stroke.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service d'Anesthésie - Réanimation, CHU Angers, Angers
  - Service d'Anesthésie - Réanimation, Groupe Hospitalier Pellegrin CHU de Bordeaux, Bordeaux
  - Service de Réanimation - CH Annecy Genevois, Epagny METZ Tessy
  - Service d'Anesthésie - Réanimation, Hôpital Michallon- CHU Grenoble, La Tronche
  - Service d'Anesthésie - Réanimation, HCL Edouard Herriot, Lyon
  - Service d'Anesthésie-Réanimation, HCL Lyon Sud, Pierre-Benité
  - Service d'Anesthésie - Réanimation, HIA St Anne Toulon, Toulon